CLINICAL TRIAL: NCT00469807
Title: Maternal Serum Ghrelin Levels in Early IVF Pregnancies: Lack of Prognostic Value for Gestational Outcome and Altered Post-Prandial Responses
Brief Title: Ghrelin Levels in Early IVF Pregnancies
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Other Study IDs: VLC-CV-0604-507-22
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy
Keywords: Ghrelin; Pregnancy outcome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, we have assessed the potential prognostic value for gestational outcome of maternal ghrelin levels at very early stages of IVF pregnancies. In addition, ghrelin responses to meal intake were explored at early gestation.

DETAILED DESCRIPTION:
Ghrelin is a pleiotropic hormone recently involved in the control of growth and metabolism, whose circulating levels fluctuate in relation to food intake and body mass index. Ghrelin has been detected in the decidualized endometrium, as well as in human and rat placenta, with a distinctive temporal pattern of expression along pregnancy.

Comparison(s): A total of 106 patients undergoing IVF procedures were prospectively recruited. On d-16 and 23 after oocyte retrieval, the patients were subjected to blood sampling after overnight fasting, for determination of serum ghrelin, hCG and progesterone levels. In addition, ghrelin levels were assayed in these groups, 2-h after ingestion of a fixed-calorie meal.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-06; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, MD, Study Chair — Instituto Valenciano de Infertilidad
Locations (1):
- Ivi Valencia, Valencia, Spain